CLINICAL TRIAL: NCT06721533
Title: Cerebellar Metaplasticity in the Swallowing Motor System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Ayodele Sasegbon, Dr, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 341596
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Swallowing; Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Arm 1 (Experimental): 1. Real 10 Hz cerebellar rTMS (250 pulses) to the right cerebellar hemisphere immediately followed by 1 Hz cerebellar rTMS (600 pulses) to the same area. Pharyngeal motor evoked potential (PMEP) amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 2 (Experimental): 2. Sham 10 Hz cerebellar rTMS (250 pulses) to the right cerebellar hemisphere immediately followed by 1 Hz cerebellar rTMS (600 pulses) to the same area. PMEP amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 3 (Experimental): 3. Real 10 Hz cerebellar rTMS (250 pulses) to the right cerebellar hemisphere followed after 45 minutes by 1 Hz cerebellar rTMS (600 pulses) to the same area. PMEP amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 4 (Experimental): 4. Real 10 Hz cerebellar rTMS (250 pulses) to the right cerebellar hemisphere followed after 90 minutes by 1 Hz cerebellar rTMS (600 pulses) to the same area. PMEP amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 5 (Experimental): 5. Real 1 Hz cerebellar rTMS (600 pulses) to the right cerebellar hemisphere immediately followed by 10 Hz cerebellar rTMS (250 pulses) to the same area. PMEP amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 6 (Experimental): 6. Sham 1 Hz cerebellar rTMS (600 pulses) to the right cerebellar hemisphere immediately followed by 10 Hz cerebellar rTMS (250 pulses) to the same area. PMEP amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 7 (Experimental): 7. Real 1 Hz cerebellar rTMS (600 pulses) to the right cerebellar hemisphere followed after 30 minutes by 10 Hz cerebellar rTMS (250 pulses) to the same area. PMEP amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 8 (Experimental): 8. Real 1 Hz cerebellar rTMS (600 pulses) to the right cerebellar hemisphere followed after 60 minutes by 10 Hz cerebellar rTMS (250 pulses) to the same area. PMEP amplitude measured
  Interventions: Device: Cerebellar rTMS
- Arm 9 (Experimental): Most excitatory metaplastic protocol (comparing effects of arms 1-8 against one another) to right cerebellar hemisphere. Swallowing accuracy measurements.
  Interventions: Device: Cerebellar rTMS
- Arm 10 (Experimental): Single dose cerebellar rTMS to right hemisphere. Swallowing accuracy measurements.
  Interventions: Device: Cerebellar rTMS

INTERVENTIONS:
Device: Cerebellar rTMS — Cerebellar rTMS applied to pharyngeal area of right hemisphere

SUMMARY:
Dysphagia is common and leads to significant morbidity and mortality within healthcare settings. Current approaches to dysphagia management involve altering the consistency of food and fluids. However, these approaches are not supported by a robust evidence base. Repetitive transcranial magnetic stimulation (rTMS) offers a non-invasive way to manipulate neuroelectric activity within the brain. Within the swallowing motor system, rTMS at a frequency of 5Hertz (Hz) and above is excitatory while 1Hz is suppressive.

Cortical rTMS targeting pharyngeal motor areas can alter brain activity and swallowing behaviour in healthy participants and has been shown to improve post-stroke dysphagia (PSD). Despite this, it has a small seizure risk. Cerebellar rTMS is a newer and safer technique which is more easily targeted and is effective at altering swallowing related brain activity and behaviour. Recent studies have also shown it can improve PSD.

Critically, individual responsiveness to rTMS is variable, potentially reducing its effectiveness. Metaplasticity whereby the brain is preconditioned with a neuroelectric stimulus before the treating stimulus is administered is a potential way of reducing variability. Metaplasticity has recently been shown to improve responses within the swallowing motor system following cortical rTMS. However, to date no cerebellar rTMS study has applied this approach. This is a gap in our understanding which will need to be addressed.

The overarching aim of the study is to develop a less variable and more effective treatment for neurogenic dysphagia. More specifically the study objectives are to establish:

1. Whether 10Hz Cer-rTMS delivered over hemispheric pharyngeal areas can induce SMS metaplastic changes in healthy participants.
2. If a cerebellar rTMS metaplastic stimulation protocol can affect swallowing behaviour.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants > 18 years of age

Exclusion Criteria:

Exclusion criteria will be the presence or a history of:

1. Epilepsy
2. Cardiac pacemaker
3. Previous brain surgery
4. Previous swallowing problems
5. The use of medication which acts on the central nervous system
6. Any implanted metal in the head
7. Pregnancy (self-declared)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Pharyngeal motor evoked potential (PMEP) amplitude | 10 measurements made at baseline, 0 minutes post stimulation, 15 minutes post stimulation, 30 minutes post stimulation, 45 minutes post stimulation and 60 minutes post stimulation
  PMEP amplitude measured using single pulse transcranial magnetic stimulation over pharyngeal motor areas of the cortex and cerebellum
Swallowing accuracy | 10 measurements made at baseline, 0 minutes post stimulation, 15 minutes post stimulation, 30 minutes post stimulation, 45 minutes post stimulation and 60 minutes post stimulation
  Swallowing accuracy measured using a reaction time task

CONTACTS AND LOCATIONS:
Overall Officials: Ayodele Sasegbon, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: No
No identifiable data pertaining to individual participants will be shared with other researchers